CLINICAL TRIAL: NCT02053441
Title: The Efficacy of Leucine Enriched-EAA Supplements vs. Whey Protein in the Modulation of Muscle Protein Synthesis, Albumin Synthesis and Leg/ Muscle Blood Flow in Older Women
Brief Title: Modulation of Muscle Protein Synthesis With Diet and Exercise in Old Aged Women
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Syed Bukhari, Research Student, University of Nottingham
Other Study IDs: C14082012
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Sarcopenia
Keywords: Muscle Protein Synthesis; Muscle Protein Breakdown
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for Glucose and RNA analysis Muscle biopsies for protein synthesis
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study will measure differences in how muscle responds to both exercise and protein supplements in healthy women aged 60-69. We are studying two different protein supplements- a standard Whey Protein and a Leucine enriched supplement. Each patient would receive either one of these.

DETAILED DESCRIPTION:
One of the factors that plays an important role in the loss of functional performance and, as such, the capacity to maintain a healthy, active lifestyle is the progressive loss of skeletal muscle mass with ageing (i.e., sarcopenia). Indeed, sarcopenia is a more robust predictor of functional status and mortality in the elderly than chronological age or indeed, any other co-morbidity. Sarcopenia is an incipient process whereby lean muscle mass contributing up to ~50% of total body weight in young adults declines to ~25% when reaching the age of 75-80 y. Adequate nutritional intake, and in particular dietary protein, is important for offsetting age-related declines in muscle mass. The aim of this project is to seek the most effective nutrition with which to counteract sarcopenia, specifically in women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal females aged 60-70

Exclusion Criteria:

* • Obvious muscle wasting.

  * A body mass index (BMI) < 18 or > 40 kg•m2.
  * Active cardiovascular disease: uncontrolled high blood pressure, angina, heart failure (class III/IV), abnormal heart rhythm, right to left cardiac shunt or recent cardiac event.
  * Taking statin-based medication above 60mg•day-1.
  * Individuals taking beta-adrenergic blocking agents or Non-steroidal anti-inflammatory agents (NSAIDS)
  * Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial).
  * Respiratory disease including pulmonary hypertension, chronic obstructive pulmonary disease (COPD), asthma or a forced expiratory volume (FEV1) less than 1.5 litres.
  * Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes.
  * Active inflammatory bowel disease, renal disease, or malignancy.
  * Recent steroid treatment (within 6 months), or hormone replacement therapy.
  * Clotting dysfunction e.g. Deep vein thrombosis, pulmonary embolus, warfarin therapy and/ or haemophilia.
  * Musculoskeletal or neurological disorders.
  * Any leg amputated
  * Family history of early (<55y) death from cardiovascular disease.
  * Known sensitivity to SONOVUE (US contrast).

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy females aged 60-70
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis and muscle protein breakdown | 7 Hours
  Markers of muscle protein synthesis and breakdown are determined from muscle biopsy samples in form of myofibrillar Fractional Synthetic Rate (FSR) assessed by gas-chromatography-combustion-mass spectrometry, using incorporation of a stable isotope tracer (13-C-6 Phe)

SECONDARY OUTCOMES:
Blood flow (bulk and nutritive) and intramuscular cell signalling | 7 Hours
  1. Leg blood flow via Common femoral bulk flow (Doppler ultrasound)
  2. Microvascular blood flow via contrast enhanced ultrasound
  3. Mammalian Target of Rapamycin-1 (mTORC1) and Protein Kinase B (PKB or AKT) phosphorylation via western immunoblotting

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Smith, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham (Derby campus), Derby, Derbyshire, United Kingdom

REFERENCES:
- [Result] Wilkinson DJ, Bukhari SSI, Phillips BE, Limb MC, Cegielski J, Brook MS, Rankin D, Mitchell WK, Kobayashi H, Williams JP, Lund J, Greenhaff PL, Smith K, Atherton PJ. Effects of leucine-enriched essential amino acid and whey protein bolus dosing upon skeletal muscle protein synthesis at rest and after exercise in older women. Clin Nutr. 2018 Dec;37(6 Pt A):2011-2021. doi: 10.1016/j.clnu.2017.09.008. Epub 2017 Sep 23. PMID 29031484
- [Result] Bukhari SS, Phillips BE, Wilkinson DJ, Limb MC, Rankin D, Mitchell WK, Kobayashi H, Greenhaff PL, Smith K, Atherton PJ. Intake of low-dose leucine-rich essential amino acids stimulates muscle anabolism equivalently to bolus whey protein in older women at rest and after exercise. Am J Physiol Endocrinol Metab. 2015 Jun 15;308(12):E1056-65. doi: 10.1152/ajpendo.00481.2014. Epub 2015 Mar 31. PMID 25827594